CLINICAL TRIAL: NCT04212156
Title: Validity of Thyromental Height Test (TMHT) as an Objective Predictor of Difficult Airway in Obese Patients: a Prospective Observational Cohort Study
Brief Title: Thyromental Height Test (TMHT) as a Predictor of Difficult Airway in Obese Patients
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Ahmed, MD, Assistant Professor of Anesthesia, SICU & pain management. Kasralainy Faculty of medicine, Cairo University
Other Study IDs: Ms-266-2019
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Difficult Airway Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TMH test: Patient will be asked to lay supine while the head and neck maintained in a neutral position using a pillow under the head. By using digital depth gauge, the TMH will be measured from the anterior border of the thyroid cartilage directly on the thyroid notch till the anterior border of the mentum

SUMMARY:
Difficult airway management is a major concern for anesthetists and contributes to perioperative morbidity and mortality. The incidence of difficult intubation in the obese population with a BMI of greater than 30 has been reported to be 15.8%. Thyromental height test (TMHT) is a new bedside test for difficult airway, it is a measure of the height between the anterior borders of the mentum and thyroid cartilage. TMHT can act as a surrogate for amount of mandibular protrusion; dimensions of submandibular space; and anterior position of the larynx. It appears promising as a single anatomical measure to predict the risk of difficult laryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18-60 years old, ASA physical status II& III with BMI > 30 Kg/m2 who will undergo elective surgical procedures under general anesthesia using endotracheal intubation with conventional laryngoscopy

Exclusion Criteria:

* Patients with neuromuscular disorders, craniofacial abnormalities, abnormal dentition, uncooperative, who need awake intubation and patients who undergoing emergency operations will be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients of both sex, aged between 18-60 years old, ASA physical status II& III with BMI > 30 Kg/m2 who will undergo elective surgical procedures under general anesthesia using endotracheal intubation using conventional laryngoscopy
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
TMHT | before induction of general anesthesia
  Validity of TMHT for prediction of difficult airway in obese patient undergoing general anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Abeer Ahmed, Maadi, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided